CLINICAL TRIAL: NCT05783531
Title: AIMDiV: Accessing Innovative Mental Health Services for Depression in Vietnam
Brief Title: Accessing Innovative Mental Health Services for Depression in Vietnam
Acronym: AIMDiV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Grand Challenges Canada (Other); Ministry of Labour, Invalids and Social Affairs (MOLISA): Vietnam (Unknown)
Responsible Party: Principal Investigator, John O'Neil, Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFU ORS 26172; R-TTS-2205-52454 (Other Grant/Funding Number: Grand Challenges Canada)
Record Dates: First submitted 2023-03-08; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Depression; Anxiety Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will receive the VMood digital mental health intervention. This consists of bibliotherapy that is delivered via a smartphone app, with coaching support provided by social workers for a duration of three months. The skills in the workbook are grounded in principles of Cognitive Behavioural Therapy.
  Interventions: Other: VMood
- Control (Other): This arm will receive enhanced treatment as usual, which consists of regular care as provided by primary care centres and a brief introduction video about depression via the app. The control arm will receive the intervention after the intervention arm has completed the intervention period.
  Interventions: Other: Enhanced treatment as usual

INTERVENTIONS:
Other: VMood — VMood is a digital mental health intervention adapted from an evidence-based in-person intervention. It uses supported self-management approaches, consisting of bibliotherapy (the Antidepressant Skills Workbook) and supportive coaching from a social worker that are provided via the smartphone app. The individual is supported in the use of the skills over the course of three months. The skills in the workbook are grounded in principles of Cognitive Behavioural Therapy.
  Arms: Intervention
Other: Enhanced treatment as usual — Participants in the control arm will receive enhanced treatment as usual in the form of usual care from primary care centres and a brief introduction to depression video through the VMood app.
  Arms: Control

SUMMARY:
This stepped wedge, randomized controlled trial (RCT) will test the effectiveness of a digital mental health intervention (VMood) adapted from an evidence-based in-person intervention. The in-person intervention is based on principles of Cognitive Behavioural Therapy and uses a supported self-management approach consisting of a patient skills workbook and supportive coaching by a non-specialist provider. It was developed in Canada and shown to be effective in the Vietnamese context in a previous RCT conducted by the research team. The digital adaptation (VMood) is delivered via a Smartphone app the research team developed in Vietnam, in close collaboration with the Institute of Population, Health and Development (PHAD) in Vietnam.

The digital intervention will be delivered at the community level in 8 Vietnamese provinces, with remote coaching provided via the app by social workers. The primary outcome measure for the study is the Patient Health Questionnaire (PHQ-9), which screens for depression caseness. The investigators will also include the Generalized Anxiety Disorder(GAD-7) measure, as symptoms of anxiety commonly co-occur with depression. Secondary outcome measures will include the WHO Quality of Life-Brief (WHOQUAL-BREV), FAST Alcohol Screening Test (FAST), the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) adapted to assess tobacco use only. The investigators will also conduct a cost-effectiveness analysis (CEA) using the 5-level EQ-5D (EQ-5D-5L), the Health Economic Assessment (HEA) adapted for the Vietnamese health context, and Work Productivity and Activity Impairment Questionnaire: Depression (WPAID:D). Finally, the System Usability Scale (SUS) will be used to assess VMood usability.

ELIGIBILITY:
Inclusion Criteria:

* Score of >4 on PHQ-9 indicating depression caseness
* consent to participate and complete all measures

Exclusion Criteria:

* Cognitive disturbance
* Psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) - change in depression scores | Monthly from baseline until three months, with a follow-up at six months
  A brief (9-item) measure for diagnosing and measuring severity of depression
Generalized Anxiety Disorder (GAD-7) - change in anxiety scores | Monthly from baseline until three months, with a follow-up at six months
  A brief (7-item) measure for assessing generalized anxiety disorder

SECONDARY OUTCOMES:
WHO Quality of Life- Brief (WHOQOL-BREV) | Three months, with a follow up at six months
  To measure the effect of the intervention on quality of life
Fast Alcohol Screening Test (FAST) | Three months, with a follow up at six months
  To measure changes in the use of alcohol products
Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) - Adapted | Three months, with a follow up at six months
  To measure changes in the use of tobacco products

OTHER OUTCOMES:
EQ-5D-5L | Three months, with a follow up at six months
  For cost-effectiveness analysis; to estimate health-related quality of life
Health Economic Assessment (HEA) - Adapted | Three months, with a follow up at six months
  For cost-effectiveness analysis; to estimate costs attributable to health resource utilization
Work Productivity and Activity Impairment Questionnaire: Depression (WPAID:D) | Three months, with a follow up at six months
  For cost-effectiveness analysis; to measure indirect costs attributable to potential productivity gains
System Usability Scale (SUS) | Three months, with a follow up at six months
  To assess the usability of the VMood app. The System Usability Scale (SUS) is an industry standard, validated 10-item Likert-type scale with five response options for measuring usability with 0 (strongly disagree) to 4 (strongly agree). Item scores are summed and the total is multiplied by 2.5. The composite score (between 0 and 100) provides an indicator of perceived usability - a higher score means better perceived ease of use. Research shows a score >68 is considered above average. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.

REFERENCES:
- [Derived] Chau LW, Murphy JK, Nguyen VC, Xie H, Lam RW, Minas H, Zheng Y, Krebs E, Hayashi K, Dao S, Nguyen X, Duong VA, Fiume E, O'Neil J. Evaluating the effectiveness and cost-effectiveness of a digital, app-based intervention for depression (VMood) in community-based settings in Vietnam: Protocol for a stepped-wedge randomized controlled trial. PLoS One. 2023 Sep 5;18(9):e0290328. doi: 10.1371/journal.pone.0290328. eCollection 2023. PMID 37669289